CLINICAL TRIAL: NCT06565104
Title: Adding Sleep to the BWell4Life Diet and Physical Activity Intervention for Cardiometabolic Health Promotion: The Sleep2BWell Community-Based, Cluster-Randomized Trial
Brief Title: The Sleep2BWell Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Nour Makarem, PhD, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU9042; 3P50MD017341-03S2 (NIH)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Blood Pressure; Sleep Health; Diet, Healthy; Physical Activity; Weight Loss
MeSH Terms: conditions — Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BWell4Life Control Arm (Active Comparator): BWell4Life is a 4-week community health promotion program focused on lifestyle change through consumption of a healthy diet and being physically active through weekly educational sessions, setting specific, measurable, attainable, realistic, and timely (S.M.A.R.T.) goals for health behavior modification, and didactic content based on the American Heart Association (AHA) Life's Essential 8 framework. The two diet sessions include an overview of nutrition basics, examples of healthy dietary patterns and cooking methods to increase consumption of plant-based foods and healthy proteins and reduce intakes of red and processed meats, sugary foods, and sugar-sweetened beverages. The two physical activity sessions provide an overview of the physical activity guidelines and include 30-60 minutes of exercise. These sessions also address achieving and maintaining a healthy body weight. Participants will receive a Fitbit for self-monitoring and collecting sleep health and physical activity data.
  Interventions: Behavioral: Healthy Diet Sessions; Behavioral: Physical Activity Sessions
- Sleep2BWell Intervention Arm (Experimental): Sleep2BWell is a 6-week program, which consists of the 4-wk BWell4Life program enhanced with two sleep health education and group coaching sessions and addressing structural barriers to healthy sleep in NYC (light, noise, and indoor air pollution). The sleep health education sessions will incorporate didactic content, engaging animated videos, group coaching, and an interactive Q&A period. These sessions will incorporate techniques to establish regular bed and wake times, learn wind-down and wake-up routines, cope with stress through muscle relaxation and mindfulness techniques, and optimize the sleep environment. Participants will self-monitor using a Fitbit and will receive additional instruction on how to maximize health benefits of self-monitoring. They will also receive a sleep mask, ear plugs, a blue light blocker, and an indoor air purifier to address barriers to healthy sleep in the sleep environment.
  Interventions: Behavioral: Multidimensional Sleep Health Sessions; Behavioral: Healthy Diet Sessions; Behavioral: Physical Activity Sessions

INTERVENTIONS:
Behavioral: Multidimensional Sleep Health Sessions — The two sleep health educational sessions will include didactic content on defining sleep health, reviewing sleep recommendations, outlining the role of sleep in preserving cardiometabolic health, and correcting unhelpful sleep-related beliefs and debunking myths. Participants will learn to maximize the benefits of self-monitoring using a Fitbit and will receive a sleep mask, ear plugs, a blue light blocker, and an indoor air purifier to improve their sleep environment.
  Arms: Sleep2BWell Intervention Arm
Behavioral: Healthy Diet Sessions — The two diet sessions include an overview of nutrition basics, examples of healthy dietary patterns and cooking methods to increase consumption of plant-based foods such as fruits, vegetables, and whole grains, promote choosing more lean proteins such as fish, and reduce intakes of red and processed meats, sugary foods, and sugar-sweetened beverages.
Behavioral: Physical Activity Sessions — The two physical activity sessions provide an overview of the physical activity guidelines and include 30-60 minutes of exercise and a healthy living community resource mapping exercise. These sessions also address achieving and maintaining a healthy body weight.

SUMMARY:
Improving multiple domains of cardiometabolic health (CMH) through contextual behavioral interventions has the potential to substantially reduce persistent chronic disease disparities. Sleep is critical for preserving CMH and is amenable to intervention in real-world settings. Although sleep health, in conjunction with other lifestyle behaviors, can improve CMH through complementary or synergistic pathways, most existing lifestyle change programs focus solely on diet and physical activity. Sleep2BWell is a community-based cluster randomized trial aimed at evaluating the impact of incorporating a multidimensional sleep health intervention into the BWell4Life program, an ongoing 4-week program for promoting CMH through healthy diet and physical activity, delivered by peer health educators at faith-based organizations and community centers in underserved NYC neighborhoods. The enhanced 6-week intervention, Sleep2BWell, will include the following additional components: 1) two sleep health education and group coaching sessions, 2) self-monitoring and motivational enhancement using a Fitbit, and 3) addressing prevalent environmental barriers to healthy sleep in urban settings such as noise and light with a novel and timely extension to address indoor air pollution. A total of 14 community sites will be randomized into the intervention (Sleep2BWell) or control (BWell4Life) group, enrolling an average of 15 participants per site for an expected sample of 210. The investigators will collect objective measures of sleep and physical activity throughout the study, and assess diet and CMH outcomes at baseline, 10 weeks (primary endpoint), and 24 weeks (long-term follow-up to assess sustainability of the intervention's effect). The investigators hypothesize that Sleep2BWell will enhance the effectiveness of BWell4Life leading to greater improvements in CMH, including reduced blood pressure (primary outcome) improved health behaviors (sleep, diet, physical activity) and adiposity markers (secondary outcomes), as well as better glycemic control and inflammatory and allostatic load indicators (exploratory outcomes). To ensure the successful completion and future expansion of this work, this study will use mixed methods to understand implementation determinants and outcomes, guided by implementation science frameworks. This first-of-its-kind effectiveness-implementation study, addressing individual level behaviors and factors and upstream influences and leveraging key behavior change and community engagement strategies, will investigate the integration of sleep health into a multi-behavior lifestyle change intervention aimed at addressing CMH disparities in community settings. This innovative multilevel intervention will inform scalable sustainable community health approaches and public health policy to improve sleep health and CMH disparities through advancement in novel multilevel bundled behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

1. English- and/or Spanish-speaking
2. aged ≥20 years
3. having at minimum SBP in the elevated or hypertension category (i.e., SBP ≥120 mmHg)

Exclusion Criteria:

1. No known medical conditions that would prevent them from safely participating in the trial (e.g., neurological degenerative disease such as Parkinsons, severe psychiatric disorders, substance use disorder)
2. History of cardiovascular disease or cancer
3. Pregnant or desire to become pregnant during the study
4. Less than one year postpartum

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | baseline to 10 weeks
  The change systolic blood pressure (mmHg) from baseline to follow-up at 10 weeks will be calculated and compared across randomization arms.

SECONDARY OUTCOMES:
Change in systolic blood pressure (sustained effect at 24 weeks) | baseline, 24 weeks
  The change in systolic blood pressure (mmHg) from baseline to follow-up at 24 weeks will be calculated and compared across randomization arms.
Change in diastolic blood pressure | baseline, 10 weeks, 24 weeks
  The change diastolic blood pressure (mmHg) from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep health | baseline, 10 weeks, 24 weeks
  Sleep health will be assessed using sleep duration, regularity, efficiency, and timing from the Fitbit and self-reported sleep satisfaction and alertness (measured by daytime sleepiness). Optimal sleep health will be defined as having an average sleep duration (hours/night) ≥7 hours and <9 hours, regular sleep duration and timing (standard deviation of sleep duration and timing variables <90 minutes), sleep efficiency (%) ≥85%, an earlier sleep period (sleep midpoint earlier than 4:00 AM), normal daytime sleepiness (Epworth Sleepiness Scale ≤10), and good self-rated sleep satisfaction and quality. Sleep health will be assessed at baseline, 10 weeks, and 24 weeks. Changes in sleep health from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep duration | baseline, 10 weeks, 24 weeks
  Sleep duration (hours) will be assessed at baseline, 10 weeks, and 24 weeks. Changes in sleep duration from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep efficiency | baseline, 10 weeks, 24 weeks
  Sleep efficiency (%) will be assessed at baseline, 10 weeks, and 24 weeks. Changes in sleep efficiency from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep regularity | baseline, 10 weeks, 24 weeks
  Sleep regularity will be assessed from the standard deviation of sleep duration and timing at baseline, 10 weeks, and 24 weeks. Changes in sleep regularity from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep quality | baseline, 10 weeks, 24 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (score range: 0-21) at baseline, 10 weeks, and 24 weeks. Changes in sleep quality from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in alertness | baseline, 10 weeks, 24 weeks
  Alertness will be captured by measuring excessive daytime sleepiness using the Epworth Sleepiness Scale (range: 0-24) at baseline, 10 weeks, and 24 weeks. Changes in daytime sleepiness from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in diet quality | baseline, 10 weeks, 24 weeks
  The change in the Mediterranean Eating Pattern for Americans (MEPA) score (range: 0-16 with higher scores indicating more favorable diet quality) from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in physical activity | baseline, 10 weeks, 24 weeks
  The change in minutes/week spent in moderate-to-vigorous intensity and light intensity physical activity from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in body weight | baseline, 10 weeks, 24 weeks
  The change in body weight (in lbs) from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in waist circumference | baseline, 10 weeks, 24 weeks
  The change in waist circumference (inches) from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in percent body fat | baseline, 10 weeks, 24 weeks
  The change in % body fat from baseline to follow-up at 10 weeks and 24 weeks will be calculated and compared across randomization arms.
Acceptability of Implementation | 10 weeks
  Acceptability will be measured by questionnaire. Items are adapted from the validated Acceptability of Implementation Measure (AIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better intervention acceptability. The items are analyzed individually and not summed to a total score.
Feasibility of Implementation | 10 weeks
  Feasibility will be measured by questionnaire using items adapted from the validated Feasibility of Implementation Measure (FIM) and rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better feasibility. The items are analyzed individually and not summed to a total score.
Appropriateness of Implementation | 10 weeks
  Appropriateness will be measured by questionnaire. Items are adapted from the validated Implementation Appropriateness Measure (IAM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better appropriateness. The items are analyzed individually and not summed to a total score.

OTHER OUTCOMES:
Change in fasting glucose | baseline, 24 weeks
  The change in fasting glucose (mg/dl) from baseline to follow-up at 24 weeks will be calculated and compared across randomization arms.
Change in allostatic load | baseline, 24 weeks
  Allostatic load will be measured by cardiovascular system, metabolic system, and inflammatory/immune system markers. Allostatic load will be computed such as that a score of 1 is assigned when a biomarker falls at or above a defined threshold (high risk) and a score of 0 is assigned when a biomarker falls below a defined threshold (low risk). High-risk thresholds are based on the following clinically defined cut points: 1) systolic blood pressure ≥140 mmHG, 2) diastolic blood pressure ≥90 mmHG, 3) total cholesterol ≥240 mg/dL, 4) HDL cholesterol <50 mg/dL, 5) triglycerides ≥150 mg/dL, 6) BMI >30.0 kg/m2, 7) waist-to-hip ratio >0.85, 8) HbA1c ≥5.5%, 9) CRP >3.0 μg/dL, and 10) IL-6 >6.5 pg/mL. The total score will range from 0 to 10 with greater values indicating higher allostatic load. The change in allostatic load from baseline to 24 weeks will be calculated and compared across randomization arms.
Change in total cholesterol | baseline, 24 weeks
  The change in total cholesterol (mg/dL) from baseline to 24 weeks will be calculated and compared across the randomization arms.
The change in HDL cholesterol | baseline, 24 weeks
  The change in HDL cholesterol (mg/dL) from baseline to 24 weeks will be calculated and compared across the randomization arms.
The change in triglyceride levels | baseline, 24 weeks
  The change in triglyceride levels (mg/dL) from baseline to 24 weeks will be calculated and compared across the randomization arms.
The change in C-Reactive Protein (CRP) levels | baseline, 24 weeks
  The change in CRP levels (μg/dL) from baseline to 24 weeks will be calculated and compared across the randomization arms.
The change in Interleuken-6 (IL-6) levels | baseline, 24 weeks
  The change in CRP levels (pg/mL) from baseline to 24 weeks will be calculated and compared across the randomization arms.

CONTACTS AND LOCATIONS:
Overall Officials: Nour Makarem, PhD, FAHA, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - Columbia University Irving Medical Center, Mailman School of Public Health, New York, New York

IPD SHARING:
Plan to Share IPD: No
Data will be shared consistent with guidance from NIMHD-funded HEAN coordinating center.